CLINICAL TRIAL: NCT03084744
Title: Senzoku Intervention of Schema Therapy for Aid and Recovery From Chronic Depression (SISTAR*CD)
Brief Title: Schema Therapy for Chronic Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Health Economics and Policy, Japan (Other)
Collaborators: Senzoku Stress Coping Support Office (Unknown)
Responsible Party: Principal Investigator, Yasuyuki Okumura, Principal Investigator, Institute for Health Economics and Policy, Japan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16207
Record Dates: First submitted 2017-03-02; First posted 2017-03-21 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Chronic Depressive Disorder; Dysthymic Disorder
MeSH Terms: conditions — Dysthymic Disorder | interventions — Schema Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated into two groups using a web-based central allocation system. This system will confirm allocation concealment and random sequence generation.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors of the primary outcome will be blinded to treatment assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Schema therapy (Experimental): Schema therapy in an individual format will be implemented by clinical psychologists. The treatment period will be 2 years with biweekly 50-minute sessions (up to 48 sessions).
  Interventions: Behavioral: Schema therapy
- Active monitoring (Placebo Comparator): Active monitoring by telephone will be implemented by clinical psychologists. The treatment period will be 2 years with monthly 10-minute sessions (up to 24 sessions).
  Interventions: Behavioral: Active monitoring

INTERVENTIONS:
Behavioral: Schema therapy — Schema therapy for chronic depression, a face-to-face psychological intervention by clinical psychologists.
  Arms: Schema therapy
Behavioral: Active monitoring — Active tele-monitoring by clinical psychologists.
  Arms: Active monitoring

SUMMARY:
To compare the efficacy of schema therapy versus active monitoring for women with chronic depression receiving psychiatric care.

DETAILED DESCRIPTION:
A randomized, assessor-blind, single center, superiority trial will be conducted. Participants will be referred to clinical psychologists in a private counseling office (Senzoku Stress Coping Support Office, in Japan). Eligible participants will be women with chronic depression receiving psychiatric care. Participants will receive schema therapy or active monitoring during 2 years. Primary outcome will be treatment response. A total sample size of 64 (32 in each group) would be required to provide 80% power at a 2-sided significance level of 5% to detect a risk difference of 35% (response rate: 55% for schema therapy vs. 20% for active monitoring), assuming a dropout rate of 10%.

ELIGIBILITY:
Inclusion Criteria:

* Persistent depressive disorder including chronic major depressive disorder and dysthymic disorder assessed by the Structured Clinical Interview for DSM
* Scores of at least 14 on the GRID-HAMD
* Psychiatric treatment duration for depression of at least 3 years

Exclusion Criteria:

* Psychiatric hospitalization within 30 days prior to the enrollment
* Ineligible to receive the protocol treatment during 2 years
* Schizophrenia
* Bipolar disorders
* Intellectual disabilities
* Neurocognitive disorders
* Substance-related disorders

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2017-08-21 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Treatment response (% change from baseline to at 104 weeks) | Baseline, 104 weeks
  Treatment response was defined as 50% or greater reduction in depressive symptoms (the 17-item GRID-Hamilton Depression Rating Scale; GRID-HAMD) at 104 weeks compared with baseline. The GRID-HAMD will be administered by clinical psychologists who will be blinded to treatment assignments.

SECONDARY OUTCOMES:
Remission | 104 weeks
  Remission was defined as the 17-item GRID-HAMD score of 7 or less at 104 weeks.
Change in observer-rated depression severity (17-item HAMD) | Baseline, 26 weeks, 52 weeks, 78 weeks, 104 weeks
  Change in observer-rated depression severity was defined as the change score of the 17-item GRID-HAMD from baseline through 104 weeks.
Change in observer-rated depression severity (24-item HAMD) | Baseline, 26 weeks, 52 weeks, 78 weeks, 104 weeks
  Change in observer-rated depression severity was defined as the change score of the 24-item GRID-HAMD from baseline through 104 weeks. The 24-item GRID-HAMD will be administered by clinical psychologists who will be blinded to treatment assignments.
Change in self-rated depression severity | Baseline, 52 weeks, 104 weeks
  Change in self-rated depression severity was defined as the change score of the Beck Depression Scale-II (BDI-II) from baseline through 104 weeks.
Change in self-rated quality of life | Baseline, 52 weeks, 104 weeks
  Change in self-rated quality of life was defined as the change score of the EQ-5D-5L.
Medical costs | baseline through 104 weeks (assessed at each session)
  The cumulative medical costs during 104 weeks for the utilization of medical services will be assessed at each session.

CONTACTS AND LOCATIONS:
Overall Officials: Yasuyuki Okumura, PhD, Principal Investigator — Institute for Health Economics and Policy; Emi Ito, PhD, Principal Investigator — Senzoku Stress Coping Support Office
Locations (1):
- Senzoku stress coping support office, Tokyo, Ota-ku, Japan

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researchers within 3 years after the publication of the primary paper.